CLINICAL TRIAL: NCT01408992
Title: The Evaluation of Thai-version Five Minute Hearing Test to Screen Hearing in Community
Brief Title: Thai-version Five Minute Hearing Test
Acronym: Thai_FMHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Kwanchanok Yimtae, M.D., Assoc. Prof. Kwanchanok Yimtae, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: HE541135
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Hearing Loss
Keywords: Hearing screening; Questionnaire; Hearing disability
MeSH Terms: conditions — Hearing Loss | interventions — Hearing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- FMHT (Experimental): All community people will be interviewed with Thai Five Minute Hearing Test questionnaire and will be tested with an audiometry.
  Interventions: Procedure: Audiometry; Other: Thai-Five Minute Hearing Test

INTERVENTIONS:
Procedure: Audiometry — Standard hearing test performed by audiologists
Other: Thai-Five Minute Hearing Test — All subjects will be interviewed with Thai-Five Minute Hearing Test

SUMMARY:
This study is aimed to test the sensitivity and specificity of Thai-version Five Minutes Hearing test against the audiometry to screen hearing problem in community.

DETAILED DESCRIPTION:
Study Population Phu Wieng district, Khon Kaen Province was chose to be a represent of rural community in Thailand. 551 subjects were desired to cover 80% sensitivity of the original test, at 95% confidence level, 80% power, and 7% margin of error. Regarding to 22.7% of the estimated prevalence of hearing loss and 10% drop out rate, then the total subjects need was 606 persons. Subjects were divided to recruit from simple random villages, one from the municipal and the other from non-municipal area. All people in target villages whether having ear problem or not, who was older than 18 years old, could read or understand Thai language, and wanted to participate, were persuaded. Those who had aphasia, or severe mental disability, or other conditions that could not perform audiometry were excluded.

Study Procedure After consenting to participate, subjects were interviewed with Thai-FMHT. Then the subjects were undergone the audiometry in the soundproof booth performed by audiologists who were blinded the result of Thai-FMHT. Pure tone threshold at 250, 500, 1000, 2000, 3000, 4000, 6000, 8000 Hz of both ears were recorded. Tympanogram was done to confirm middle ear pathology. Any pure tone air-conduction threshold greater than 25 dB in one or two frequencies was considered as abnormal hearing. However, the severity of hearing loss was defined by pure tone average air-conduction threshold according to ASHA criteria. To compare with the original FMHT, the pure tone average air-conduction threshold at 500, 1000, and 2000 Hz was defined as speech PTA (SF-PTA), whereas, the pure tone average air-conduction threshold at 3000, 4000, 6000, 8000 Hz was defined as high frequency PTA (HF-PTA). Hearing disability was classified according to the hearing level of the better hearing ear.

Otolaryngologists did history taking. Ear symptoms such as otalgia, itching, otorrhea, tinnitus, and hearing loss was asked before performing otoscopy and making a final diagnosis. The treatment, or medication if needed, and advice were complementary provided to subjects as post-trial benefits.

Statistical analysis Descriptive analysis was used to present demographic data. The sensitivity, specificity, and ROC were analyzed using STATA software version 10.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older

Exclusion Criteria:

* having aphasia, or severe mental disability, or other conditions which can not accommodate audiometry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwanchanok Yimtae, M.D., Principal Investigator — Khon Kaen University; Pornthep Kasemsiri, M.D., Principal Investigator — Khon Kaen University; Panida Thanawirattananit, M.A., Principal Investigator — Khon Kaen University
Locations (1):
- Phu Weng, Ban Phu Wang, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Yimtae K, Kasemsiri P, Thanawirattananit P, Siripaopradith P. Validation of the Thai five-minute hearing test to screen hearing loss in the community. Audiol Neurootol. 2014;19(2):127-34. doi: 10.1159/000357492. Epub 2014 Jan 22. PMID 24457423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2011 through September 2011, 643 Eligible persons agreed to participate. 85 persons withdrew later and 558 persons complete all study procedures.
Pre-assignment Details: A total of 551 subjects were required to obtain an 80% sensitivity rate for the original test, at a 95% confidence level, with 80% power, and a 7% margin of error. Considering 22.7% as the estimated prevalence of hearing loss [Prasansuk, 2000] and a 10% drop out rate, the total number of subjects needed was 606.
Groups:
- Community People: The Phu Wieng district in Khon Kaen Province was chosen as a representative rural community in Thailand. This district comprises 114 villages and has a population of 24,201 inhabitants. Of these, 13,001 inhabitants lived in municipal areas, whereas the rest lived in non-municipal areas. The subjects were recruited from different target villages. The villages had been divided according to their municipality. The target villages were simply randomly selected from a list of villages that have more than 300 adults in their populations. One village was from a municipal area and the other village was from a non-municipal area. All of the people in the target villages, who were older than 18 years, could read or understand the Thai language, and wanted to participate, were recruited. Those who had aphasia, severe mental disability, or other conditions that precluded audiometry were excluded.
Period: Overall Study
Arm/Group | Community People
Started | 558
Completed | 558
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Community People: The Phu Wieng district in Khon Kaen Province was chosen as a representative rural community in Thailand. A total of 551 subjects were required to obtain an 80% sensitivity rate for the original test, at a 95% confidence level, with 80% power, and a 7% margin of error. Considering 22.7% as the estimated prevalence of hearing loss [Prasansuk, 2000] and a 10% drop out rate, the total number of subjects needed was 606. The subjects were recruited from different target villages. The villages had been divided according to their municipality. The target villages were simply randomly selected from a list of villages that have more than 300 adults in their populations. One village was from a municipal area and the other village was from a non-municipal area. All of the people in the target villages, who were older
Arm/Group | Community People
Number analyzed (Participants) | 558
Age, Customized [Number; unit: participants]
  18-19 years | 2
  Between 20 and 29 years | 40
  Between 30 and 39 years | 53
  Between 40 and 49 years | 109
  Between 50 and 59 years | 128
  Between 60 and 69 years | 123
  Between 70 and 79 years | 86
  >,= 80 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 382
  Male | 176

OUTCOME MEASURES:

1. Secondary Outcome: Prevalence of Ear Diseases
Description: the frequency of diseased ears per the total examined ears
Time Frame: Immediate
Measure: Number; unit: ears
Units Other Than Participants: ears
Groups:
- Normal Ears and Hearing: Normal ear examination and normal hearing
- Ear Wax: Impacted cerumen
- Otitis Media With Effusion: Fluid in middle ear, whether serous, mucoid, mucous, or pus
- Chronic Otitis Media: Tympanic membrane perforation with or without ear discharge
- Conductive Hearing Loss: Air-bone gap and bone conduction thresholds are lower than 25 dB
- Sensorineural Hearing Loss: Air and bone conduction thresholds are more than 25 dB
- Mixed Hearing Loss: Air and bone conduction threshold are more than 25 dB with air-bone gap
Arm/Group | Normal Ears and Hearing | Ear Wax | Otitis Media With Effusion | Chronic Otitis Media | Conductive Hearing Loss | Sensorineural Hearing Loss | Mixed Hearing Loss
Number analyzed (Participants) | 558 | 558 | 558 | 558 | 558 | 558 | 558
Number analyzed (ears) | 1116 | 1116 | 1116 | 1116 | 1116 | 1116 | 1116
ears | 497 | 144 | 3 | 12 | 14 | 587 | 19

2. Post Hoc Outcome: Sensitivity of FMHT to Detect the Hearing Loss.
Description: FMHT has 15 questions and there are 4 possible answer for each question. The best possible answer is "never" and is scored "0", "occasionally" is scored "1", "half the time" is scored "2" and "almost always" the worst answer is scored "3". The total possible range for the FMHT scores 0-45. We then compared the total score with the better hearing ears as in Outcome measure 1. The total number of participants with a score from 0 to 45, and that all participants in the study had a score within this range. It would appear, from information provided in the previous version of this record, that the total score might range from 0 to 45.
Time Frame: baseline
Population: The frequencies of subjects who had FMHT score from 0 to 45 were counted.
Measure: Number; unit: participants
Groups:
- FMHT: FMHT Score is the sum of value of the answers for each question. If the subject answers "never", it will be scored as 0, "occasionally" will be 1, "half the time" will be 2, and "almost always" will be 3.
Arm/Group | FMHT
Number analyzed (Participants) | 558
participants | 558

3. Primary Outcome: Standard Hearing Test
Description: Hearing loss is defined as an elevation, at least more than 25 dB of air-conduction, pure tone average threshold at speech frequencies. The severity loss is categorized into mild (26-40 dB), moderate (41-55 dB), moderately severe (56-74 dB), severe (75-90 dB), and profound (>90 dB). In this study, we aim to use FMHT as a screening tool for hearing disability (Better hearing ear has hearing threshold greater than 40 dB).
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Hearing Loss: The severity of hearing loss was defined by the pure tone average air-conduction threshold at the speech frequencies of the better hearing ears, according to the ASHA criteria. Normal hearing means PTA of less than or equal 25 dB. Mild hearing loss means PTA of 26-40 dB. Moderate hearing loss means PTA of 41-55 dB. Moderately severe hearing loss means PTA of 56-74 dB. Severe hearing loss means PTA of 75-90 dB. Profound hearing loss means PTA > 90 dB.
Arm/Group | Hearing Loss
Number analyzed (Participants) | 558
participants
  Normal Hearing | 422
  Mild Hearing Loss | 107
  Moderate Hearing Loss | 24
  Moderately Severe Hearing Loss | 4
  Severe Hearing Loss | 1
  Profound Hearing Loss | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Community People: All people who live in the Phu Wieng district in Khon Kaen Province was chosen as a representative of community people in Thailand.
Arm/Group | Community People
Serious Adverse Events (participants affected / at risk) | 0/558
Other Adverse Events (participants affected / at risk) | 0/558

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less